



# RESEARCH PARTICIPANT INFORMED CONSENT FORM (THINK-ALOUD INTERVIEW)

Please read this document carefully before you decide to participate in this research study. Your participation is voluntary, and you can decline to participate, or withdraw consent at any time, with no consequences.

#### **Study Title:**

Adapting and Pilot Testing a Nutrition Module delivered with Virtual Human Technology for Colorectal Cancer Prevention

#### Person(s) conducting the research:

Melissa Vilaro, Postdoctoral Associate, STEM Translational Communication Center, College of Journalism and Communications, University of Florida, <a href="mailto:mgraveley@ufl.edu">mgraveley@ufl.edu</a>, (352) 846-3014

Janice Krieger, Director, STEM Translational Communication Center, College of Journalism and Communications, University of Florida, <u>Janicekrieger@ufl.edu</u>, (352) 273-0204

Ben Lok, Professor, Computer & Information Sciences & Engineering Department, University of Florida, <a href="lok@cise.ufl.edu">lok@cise.ufl.edu</a>, (352) 450-6308

## Purpose of the research study:

This study uses the opinions of adults between the ages of 50 and 73 years old to develop and test an interactive nutrition module for use in an existing colorectal cancer screening intervention using virtual human technology. This study will contribute to knowledge of what messages and graphics promote understanding of cancer risk and promote screening.

# What you will be asked to do in the study:

You will be asked to interact with an interactive web-based application (or app) containing a virtual health assistant that will talk to you about nutrition and colorectal cancer screening.

IRB Project #: 201902537 

IRB Version: 12/1/2018

You will be asked to think aloud (say whatever comes to your mind) as you interact, with the virtual health assistant application. This will include:

- Saying your thoughts about what you see (pictures, words, setting)
- Describing your feelings as you interact with the app
- Describing out loud what you are doing as you move through the app
- Detailing problems, issues, and barriers you find during the interaction
- Thinking out loud about different aspects of the app (easy to use)
- Filling out a questionnaire about yourself and experiences with the app

The interview will be audio and video recorded so that researchers can review the discussion at later dates.

## Time required:

Approximately 1 hour.

#### Risks and benefits:

There are no risks or discomforts anticipated. There are no direct benefits of participation for you. As a result of participation in the study, you may have a better understanding of your health.

#### **Confidentiality:**

Your identity will be kept confidential to the extent provided by law. Researchers will take every precaution to maintain confidentiality of the information you share. Your information will be assigned a code number. The list connecting your name to the code number will be kept in a locked file.

Your name or personal information will not be identified on the video or audio recordings, and confidentiality will be strictly maintained. However, when these video and/or audio recordings are shown or heard, the research staff may be able to identify you. Information will be kept on a password protected computer and/or an encrypted hard drive. Your name will not be used in any report.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

IRB Project #: 201902537 

IRB Version: 12/1/2018

Study ID:IRB201902537 Date Approved: 10/5/2020



#### **Compensation:**

You will be given a \$35 gift card for your participation.

## Source(s) of funding for the research:

Funding for this study is provided by National Institutes of Health (NIH) National Cancer Institute (NCI) as a supplement under award number R01CA207689-02.

#### May the researcher(s) benefit from the research?

We may benefit professionally if the results of the study are presented at meetings or in scientific journals.

#### Withdrawal from the study:

You are free to withdraw your consent and to stop participating in this study at any time without consequence. You can decline to answer any question you don't wish to answer.

#### If you withdraw, will your information be used or discarded?

Information collected will be used up until the withdrawn date/time, unless the participant requests for the data collected to not be used.

If you wish to discuss the information above or any discomforts you may experience, please ask questions now or contact one of the research team members listed at the top of this form.

If you have any questions regarding your rights as a research subject, please contact the Institutional Review Board (IRB02) office (University of Florida; PO Box 100173; Gainesville, FL 32610; (352) 392-0433 or irb2@ufl.edu.)

#### **Agreement:**

Now that you've read about the study, if you wish to participate, click the "I agree to participate" button to continue; if you do not consent to participate, click "I do not wish to participate" or just close this window.

| I agree to participat | re |
|---------------------------------------------|----------|
| I do not wish to par | ticipate |
| *If select agree to participate: | |
| Please enter your first name and last name: | |

IRB Project #: 201902537 

IRB Version: 12/1/2018

Study ID:IRB201902537 Date Approved: 10/5/2020



\*If select do not wish to participate:

Thank you!

IRB Project #: 201902537 

IRB Version: 12/1/2018